CLINICAL TRIAL: NCT07149519
Title: Impact of Dietary Guidance and Probiotics in the Treatment of Chronic Pelvic Pain Secondary to Endometriosis and Irritable Bowel Syndrome in Women: A Randomized, Double-Blind Clinical Trial
Brief Title: Impact of Dietary Guidance and Probiotics in the Treatment of Endometriosis and Irritable Bowel Syndrome in Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Letícia Lenharo, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE: 84024824.1.0000.5440
Record Dates: First submitted 2025-08-08; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Endometriosis; Bowels Irritable
Keywords: dietary; probiotics; endometriosis; bowel irritable syndrome; pelvic chronic pain
MeSH Terms: conditions — Endometriosis; Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: Specific dietary guidance associated with placebo. (Placebo Comparator): Patients in this group will receive, within 24 hours of randomization, guidance on a low-FODMAP diet, which must be followed for 12 weeks (120 days), and placebo.
  Interventions: Dietary Supplement: probiotics - Lactobacillus spp
- Arm 2: Specific dietary guidance combined with probiotics. (Experimental): Patients in this group will receive, within 24 hours of randomization, the same low-FODMAP diet guidance combined with probiotics (Lactobacillus and L. gasseri combinations) administered orally once daily for 12 weeks.
  Interventions: Dietary Supplement: probiotics - Lactobacillus spp
- Arm 3: Control - exclusive habitual diet (No Intervention): Patients in this group will be instructed to maintain their usual diet and will be administered a placebo. After the 12-week period, if the active treatment group (Arm 1 and 2) has shown a satisfactory clinical response, we will offer specific dietary guidance and probiotics to the control group participants who did not show clinical improvement.

INTERVENTIONS:
Dietary Supplement: probiotics - Lactobacillus spp — Group 1: Specific dietary guidance (low-FODMAP diet ) combined with placebo Group 2: Specific dietary guidance (low-FODMAP diet ) combined with probiotic Group 3: Control - Exclusive habitual diet After the 12-week period, we will evaluate the clinical improvement response of pelvic pain
  Other Names: Low FODMAPs dietary
  Arms: Arm 1: Specific dietary guidance associated with placebo.; Arm 2: Specific dietary guidance combined with probiotics.

SUMMARY:
Patients with endometriosis are 2 to 3 times more likely to develop Irritable Bowel Syndrome (IBS) than women without the condition. IBS presents symptoms similar to those of intestinal and deep EDT, leading to diagnostic errors and delays in identifying such comorbidities. Diets have shown positive effects on symptoms in women with both conditions, supporting the theory of a similar pathophysiology. The investigators goal is to examine how dietary practices and probiotic use affect chronic pelvic pain in patients with both comorbidities.

DETAILED DESCRIPTION:
Endometriosis (EDT) is a chronic, inflammatory, hormone-dependent disease that induces cellular adhesion and proliferation, stimulates vascularization, and disrupts protective immune responses. In its intestinal form, endometriosis can lead to abdominal pain, dyschezia, and both cyclic and non-cyclic changes in bowel habits. Patients with endometriosis are 2 to 3 times more likely to develop Irritable Bowel Syndrome (IBS) than women without the condition. IBS, which is a disorder characterized by brain-gut interactions and inflammation, presents symptoms similar to those of intestinal and deep EDT, leading to diagnostic errors and delays in identifying such comorbidities. Anti-inflammatory diets have shown positive effects on symptoms in women with both conditions, supporting the theory of a similar pathophysiology. Given the already documented alteration of the gut microbiota and the female reproductive tract, and their dysbiosis associated with the development of EDT and IBS, the investigators are encouraged to further explore the connection between them. The investigators goal is to examine how dietary practices and probiotic use affect chronic pelvic pain in patients with both comorbidities. By doing so, the investigators aim to underscore the significance of exploring non-pharmacological treatments and to provide new insights for advancing the understanding and management of endometriosis.

ELIGIBILITY:
Inclusion Criteria:

1. Women between 18 and 50 years of age who wish to participate in the clinical trial;
2. Willingness to voluntarily participate in the study and accept randomization to any of the three treatment arms;
3. Participating exclusively in this clinical trial during the study period;
4. Signing the Informed Consent Form (ICF) approved by the Research Ethics Committee (CEP) and CONEP

Exclusion Criteria:

1. Chronic, severe, or uncompensated clinical conditions, such as: malnutrition (BMI <18); insulin-dependent diabetes (types 1 or 2); uncontrolled hypertension; lung disease such as asthma or other chronic obstructive pulmonary disease; hematologic and liver diseases; advanced-stage chronic kidney disease (grades 3, 4, and 5); metabolic disorders; and immunosuppression;
2. Clinical conditions of the gastrointestinal tract that cause IBS-like symptoms, such as: inflammatory bowel disease (Chron's disease, ulcerative colitis), microscopic colitis, celiac disease, and lactose intolerance;
3. Endometriosis requiring surgical treatment during the study period;
4. Severe eating disorders, such as: bulimia, anorexia nervosa, and binge-eating disorder;
5. Chronic use of any medication with potential interaction with probiotics, the intestinal microbiota, or the natural progression of the disease in the last 6 months (such as probiotics, antibiotics, antifungals, antihistamines, digestive medications, or treatments for constipation or diarrhea);
6. Patients who already consume healthy foods or are on a restrictive diet more than four days a week, which may affect the evaluation results;
7. Patients whose stool protopastological examination is altered;
8. Inability to use oral medication;
9. Pregnancy or lactation;
10. History of alcohol or drug dependence;
11. Smoking in the last three years;
12. Inability to cooperate with investigators due to cognitive impairment or mental state.

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-02-15 (Estimated)

PRIMARY OUTCOMES:
pain improvement | 12 weeks
  visual analogic scale (EVA) EVA ranging from 0,0-10,0 Higher scores indicate worse pain.

SECONDARY OUTCOMES:
improvement in quality of life associated with bowel function | 12 week
  Gastrointestinal Quality of Live Index - GIQLI. Global score GIQLI ranging from 0-144. For the unweighted display of the global score and the dimensions, sum all item scores across the 5 domains to calculate the overall GIQLI score.
  Improvement in quality of life will be assessed by the change in the Global Score. Higher scores indicate better quality of life.
improvement of bowel function | 12 weeks
  Bristol scale. Categorizes stool consistency into seven types. Types 1 and 2 indicate constipation; types 3 and 4 are ideal stools, easy to defecate and without excess liquid; type 5 indicates a lack of fiber in the diet; and types 6 and 7 indicate diarrhea.
nutritional analysis | 12 weeks
  Food record and FODMAPS analysis by Monash University
analysis of intestinal microbiota | 12 weeks
  DNA extraction and genetic sequencing using the microway technique. Microbiota diversity will be assessed by alpha diversity (number of OTUs, Chao index) and beta diversity (weighted and unweighted UniFrac). Operational taxonomic units (OTUs) with a global abundance of less than 0.01% or presence in less than 25% of samples will be excluded from the analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Letícia Ferracini Lenharo Hayashi, Catanduva, São Paulo, Brazil